CLINICAL TRIAL: NCT02940626
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Safety and Efficacy of a Single Dose of ASN100 for the Prevention of Staphylococcus Aureus Pneumonia in Heavily Colonized, Mechanically Ventilated Subjects
Brief Title: Prevention of S. Aureus Pneumonia Study in Mechanically Ventilated Subjects Who Are Heavily Colonized With S. Aureus.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: As a result of a pre-planned interim analysis for futility
Sponsor: Arsanis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASN100-201; 2016-002146-23 (EudraCT Number)
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Pneumonia, Ventilator-associated; Pneumonia, Staphylococcal
Keywords: Pneumonia; S. aureus; Mechanically ventilated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia, Staphylococcal; Pneumonia; Staphylococcal Infections | interventions — ASN100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered as 2 separate intravenous (IV) infusions
  Interventions: Drug: Placebo
- ASN100 (Experimental): ASN100 administered as 2 separate intravenous (IV) infusions
  Interventions: Drug: ASN100

INTERVENTIONS:
Drug: ASN100 — monoclonal antibody combination of ASN-1 and ASN-2
  Other Names: ASN-1 and ASN-2
  Arms: ASN100
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is the prevention of Staphylococcus aureus pneumonia in mechanically ventilated subjects heavily colonized with S. aureus. Staphylococcus aureus is a human pathogenic bacterium that causes severe infections, including pneumonia and sepsis. Hospital-acquired bacterial pneumonia (HABP) caused by S. aureus, including ventilator-associated bacterial pneumonia (VABP) in mechanically ventilated subjects, is a significant public health threat despite efforts to optimize antibiotic treatment. ASN100 is an investigational monoclonal antibody product that targets the toxins produced by S. aureus to protect subjects from developing S. aureus pneumonia.

DETAILED DESCRIPTION:
This is a double-blind, randomized, single-dose, placebo-controlled study of ASN100 for the prevention of S. aureus pneumonia in mechanically ventilated subjects who are heavily colonized with S. aureus. This will be a global study conducted at approximately 65 sites to assess the safety, tolerability, and efficacy of ASN100.

Eligible subjects who meet all of the inclusion criteria and none of the exclusion criteria will be screened by semi-quantitative culture of an endotracheal aspirate (ETA) to identify those who are heavily colonized with S. aureus (3+ to 4+). Upon determination of eligibility, subjects will be randomized in a 1:1 ratio to 1 of 2 treatment groups, ASN100 or placebo.

ELIGIBILITY:
Inclusion Criteria:

- Subject is currently hospitalized and is mechanically ventilated endotracheally (i.e., orotracheal or nasotracheal) and, in the Investigator's opinion, will require ongoing ventilator support for at least 48 hours;

Exclusion Criteria:

* Subject has a chest X-ray or thoracic computed tomography (CT) scan that is definitive for a diagnosis of pneumonia
* Subject has a known and documented ETA culture showing heavy colonization with a -Gram-negative organism at enrollment or at any time during the Screening period;
* Significant Neutropenia
* Severe non-pulmonary source of infection.
* Subjects with a known history or current (suspected) diagnosis of cytokine release syndrome associated with the administration of peptides, proteins, and/or antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arsanis, Inc, Study Director — Arsanis, Inc.
Locations (79):
- United States (16):
  - Research Site, Phoenix, Arizona
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Chicago, Illinois
  - Research Site, Georgetown, Kentucky
  - Research Site, Hazard, Kentucky
  - Research Site, Burlington, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Buffalo, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
- Austria (2):
  - Research Site 040-001, Vienna
  - Research Site 040-002, Vienna
- Research Site, Prague, Czechia
- France (3):
  - Research Site, Argenteuil
  - Research Site, Lille
  - Research Site, Limoges
- Georgia (11):
  - Research Site 268-007, Rustavi
  - Research Site 268-005, Tbilisi
  - Research Site 268-009, Tbilisi
  - Research Site 268-004, Tbilisi
  - Research Site 268-006, Tbilisi
  - Research Site 268-002, Tbilisi
  - Research Site 268-008, Tbilisi
  - Research Site 268-011, Tbilisi
  - Research Site 268-003, Tbilisi
  - Research Site 268-010, Tbilisi
  - Research Site 268-001, Tbilisi
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Ózd
- India (6):
  - Research Site, Bangalore
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Mahara
  - Research Site, Mumbai
  - Research Site, Pune
- Israel (4):
  - Research Site, Hadera
  - Research Site, Holon
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Poland (2):
  - Research Site, Bialystok
  - Research Site, Opole
- Portugal (5):
  - Research Site, Abrantes
  - Research Site, Amadora
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Viana do Castelo
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Timișoara
- Russia (6):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Sestroretsk
- Serbia (5):
  - Research Site 688-001, Belgrade
  - Research Site 688-002, Belgrade
  - Research Site 688-005, Belgrade
  - Research Site 688-004, Kragujevac
  - Research Site 688-003, Niš
- South Africa (2):
  - Research Site, Pretoria
  - Research Site, Soweto
- Spain (6):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Tarragona
  - Research Site, Valencia
- Ukraine (4):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Lviv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized at 35 centers in the United States, Austria, Czechia, France, India, Israel, Poland, Portugal, Romania, Serbia, Spain, Rep. of Georgia, and Russian Federation
Pre-assignment Details: Eligible subjects underwent daily screening of endotracheal aspirates to determine if they met randomization criteria. Only subjects who were randomized are included in the study analysis and summarized in the Participant Flow. A single subject was randomized/treated in a site-specific pneumonia treatment sub-study.
Groups:
- ASN100: ASN100 administered as 2 separate intravenous (IV) infusions
  ASN100 3600 mg: monoclonal antibody combination of ASN-1(1800 mg) and ASN-2(1800 mg) [administered once]
- Placebo: Placebo administered as 2 separate intravenous (IV) infusions
  Placebo: Placebo [administered once]
Period: Overall Study
Arm/Group | ASN100 | Placebo
Started (Population = Intent to treat (ITT)) | 77 | 78
Randomized Into Primary Prevention Study | 77 | 77
Randomized Into Treatment Sub-study (Single subject randomized/treated (placebo) in pneumonia treatment sub-study before trial terminated) | 0 | 1
Received Study Treatment (Of the 77 subjects in the placebo arm, 76 were in primary prevention study, 1 in treatment sub-study) | 77 | 77
Completed Through Study Day 22 | 42 | 49
Completed | 30 | 43
Not Completed | 47 | 35
Not completed — Death | 40 | 32
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Transfer to Hospice Care | 1 | 0
Not completed — Prohibited Concomitant Medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: Population = Modified Intent to Treat (MITT), the population analyzed for determination of the primary endpoint. MITT includes subjects in the ITT Population who receive study drug AND who are heavily colonized with S. aureus as determined by quantitative or semi-quantitative culture of an ETA specimen prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | ASN100 | Placebo | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 43 | 83
  >=65 years | 36 | 33 | 69
Age, Continuous [Median (Full Range); unit: years] | 63.5 [24 to 92] | 62 [20 to 88] | 62.5 [20 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 50 | 50 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 70 | 71 | 141
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 71 | 74 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Romania | 1 | 2 | 3
  United States | 10 | 11 | 21
  Czechia | 1 | 0 | 1
  Portugal | 0 | 1 | 1
  India | 1 | 0 | 1
  Russia | 19 | 23 | 42
  Spain | 1 | 1 | 2
  Austria | 1 | 0 | 1
  Poland | 4 | 5 | 9
  Georgia | 34 | 29 | 63
  Israel | 1 | 3 | 4
  France | 1 | 0 | 1
  Serbia | 2 | 1 | 3
Body Mass Index Category [Mean (Standard Deviation); unit: kg/m^2] | 26.98 (5.985) | 27.17 (4.335) | 27.07 (5.209)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of a Single Intravenous (IV) Dose of ASN100
Description: Percentage of subjects in the MITT population who have or have not developed S. aureus (SA) pneumonia after a single intravenous (IV) dose of ASN100, based on sponsor defined outcome (SDO1). For each arm, the empirical proportion is defined by a ratio, which is the number of SA pneumonia events divided by the total number of subjects in the arm. The inference about the difference of two population rates is based on the empirical counterpart; specifically, the point estimate, 95% confidence interval and p-value for the rate difference. Subjects discontinued from the study due to any cause prior to Day 22 were considered as not developing SA pneumonia for the primary efficacy analysis.
Time Frame: Incidence of S. aureus pneumonia up to but not including Day 22
Population: MITT: There are 2 SDO definitions. SDO1 meets either respiratory OR signs/symptoms requirements while SDO2 must meet BOTH. Individual assessments for each randomized subject were collapsed to assign a SDO1/SDO2 of Yes, No, Indeterminate (insufficient data to assign a SDO of Yes or No), or Censored (subject died prior to the Day 22 assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | ASN100 | Placebo
Number analyzed (Participants) | 76 | 76
Participants
  Developed S. aureus Pneumonia | 5 | 7
  Did Not Develop S. aureus Pneumonia | 42 | 48
  Censored | 20 | 17
  Indeterminate | 9 | 4
Statistical Analysis 1: Comparison: ASN100 vs Placebo; Subjects were analyzed for efficacy in the group to which they randomized. Sponsor defined outcomes were based on review of microbiology results from samples tested at the central lab. If sample was not sent to the central lab., determination was based on results from the local microbiology lab. In cases where both local & central lab results were available, concordance was confirmed for S. aureus. Therefore, the analysis used local microbiology data in order to utilize a more complete dataset; Test type: Other; p = .5470, Wald Test on equality of proportions

2. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration of mechanical ventilation during the first 21 days post-randomization for subjects in the Modified Intent-to-Treat (MITT) Population
Time Frame: 21 days
Population: Modified Intent to Treat (MITT): Includes All subjects in ITT Population (randomized) who received study drug and were heavily colonized with S. aureus determined by quantitative or semi-quant. culture of an ETA specimen. Exclusion from the MITT was determined programmatically. Subjects on MV < 2 days post treatment were excluded from analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ASN100 | Placebo
Number analyzed (Participants) | 73 | 71
Days | 11.6 (7.47) | 10.1 (6.93)

3. Secondary Outcome: Length of ICU Stay
Description: Total length of ICU stay during the first 21 days post-randomization for subjects in the MITT Population
Time Frame: 21 days
Population: Modified Intent to Treat (MITT): Includes all subjects in ITT Population (randomized) who received study drug and were heavily colonized with S. aureus determined by quantitative/semi-quant. culture of an ETA specimen. Exclusion from the MITT determined programmatically. Subjects not listed as being in ICU post treatment were excluded from analysis
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ASN100 | Placebo
Number analyzed (Participants) | 74 | 75
Days | 13.7 (6.69) | 13.6 (7.21)

4. Secondary Outcome: 28-day All-cause Mortality
Description: 28-day all-cause mortality in the MITT Population
Time Frame: 28 days
Population: Modified Intent to treat (MITT): includes all subjects in the ITT Population (randomized subjects) who receive study drug and who are heavily colonized with S. aureus as determined by quantitative or semi-quantitative culture of an ETA specimen. Exclusion from the MITT Population was determined programmatically for each ITT subject.
Measure: Count of Participants; unit: Participants
Arm/Group | ASN100 | Placebo
Number analyzed (Participants) | 76 | 76
Participants | 30 | 25

5. Secondary Outcome: ASN-1 and ASN-2 Maximum Serum Concentration (Cmax)
Description: The levels of ASN-1 and ASN-2 measured at completion of study medication infusion, and at 6 hr, 24 hr, Day 4, Day 7, Day 14, Day 22, and Day 90 (final study visit) in subjects who are hospitalized or are able to return to the clinic for blood sampling.
Time Frame: through day 90
Population: Pharmacokinetic (PK) Population: All subjects in the MITT population with at least 1 serum PK sample collected post-dose. Of the 76 subjects who received ASN100, 74 were included in the PK analysis as a result of 2 not having sufficient data. Additional reductions in the number of participants analyzed is due to missing or out of window samples.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- ASN-1; ASN-2: ASN100 administered as 2 separate intravenous (IV) infusions
  ASN100: monoclonal antibody combination of ASN-1 and ASN-2. Pharmacokinetic analysis was performed and reported based on the separate antibodies (i.e. ASN-1 or ASN-2)
Arm/Group | ASN-1 | ASN-2
Number analyzed (Participants) | 71 | 73
μg/mL | 414.43 (125.55) | 460.88 (149.76)

6. Secondary Outcome: ASN-1 and ASN-2 Time to Maximum Concentration (Tmax) in Serum
Description: The levels of ASN-1 and ASN-2 measured at completion of study medication infusion, and at 6 hr, 24 hr, Day 4, Day 7, Day 14, Day 22, and Day 90 after completion
Time Frame: through day 90
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hours (from end of infusion)
Arm/Group | ASN-1 | ASN-2
Number analyzed (Participants) | 71 | 73
Hours (from end of infusion) | 6.34 (10.25) | 4.52 (5.77)

7. Secondary Outcome: ASN-1 and ASN-2 Area Under the Concentration-time Curve in Serum
Description: as for outcome 6
Time Frame: through day 90
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | ASN-1 | ASN-2
Number analyzed (Participants) | 71 | 73
μg*h/mL | 44192.3 (25080.9) | 49366.7 (29337.9)

8. Secondary Outcome: ASN-1 and ASN-2 Terminal Elimination Half-life (t1/2) in Serum
Description: as for outcome 6
Time Frame: through day 90
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ASN-1 | ASN-2
Number analyzed (Participants) | 54 | 58
Hours | 178.9 (101.13) | 185.1 (136.09)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events (AEs) analyzed include treatment-emergent AEs, from the time of randomization through the Day 90 study visit (i.e. last study visit). Only study procedure related AEs were to be reported from the time that informed consent was signed up to randomization, if they were considered to be study procedure related, however no such AEs were reported. Therefore, study procedure related AEs prior to randomization were not analyzed or reported.
Arm/Group | ASN100 | Placebo
All-Cause Mortality (participants affected / at risk) | 41/77 | 32/77
Serious Adverse Events (participants affected / at risk) | 49/77 | 38/77
Other Adverse Events (participants affected / at risk) | 74/77 | 69/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASN100 (N=77) | Placebo (N=77)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 5 (5) | 1 (1)
Cardiac Failture Acute (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Cardiovascular Insufficiency (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular Asytole (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (2)
Cardiopulmonary Failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Rupture (Cardiac disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) | 3 (3)
Death (General disorders) | 0 (0) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) — Pneumonia, which was an endpoint for the trial, was only entered as an Adverse Event (AE) if it met serious reporting criteria (i.e. SAE)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Splenic Abscess (Infections and infestations) | 1 (1) | 0 (0)
Brain Herniation (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal Shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Congestion (Nervous system disorders) | 6 (6) | 3 (3)
Brain Oedema (Nervous system disorders) | 3 (3) | 4 (4)
Coma (Nervous system disorders) | 3 (3) | 3 (3)
Ischemia Stroke (Nervous system disorders) | 3 (3) | 2 (2)
Haemorrhagic Transformation Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Nervous System Disorder (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrospinal Fluid Circulation Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 1 (1)
Deep vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Neurogenic Shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASN100 (N=77) | Placebo (N=77)
Anaemia (Blood and lymphatic system disorders) | 15 (17) | 11 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 4 (4)
Tachycardia (Cardiac disorders) | 5 (5) | 5 (6)
Tracheo-oesophageal Fistula (Congenital, familial and genetic disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 5 (7)
Pyrexia (General disorders) | 17 (25) | 8 (12)
Bronchitis (Infections and infestations) | 8 (8) | 5 (5)
Bronchitis Bacterial (Infections and infestations) | 16 (16) | 7 (7)
Sinusitis (Infections and infestations) | 4 (4) | 2 (2)
Tracheobronchitis (Infections and infestations) | 5 (7) | 7 (8)
Urinary Tract Infection (Infections and infestations) | 16 (16) | 14 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (9) | 6 (7)
Hypernatremia (Metabolism and nutrition disorders) | 5 (5) | 3 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (8) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 9 (10) | 6 (13)
Metabolic Acidosis (Metabolism and nutrition disorders) | 8 (9) | 3 (4)
Acute Kidney injury (Renal and urinary disorders) | 8 (8) | 5 (5)
Renal Failure (Renal and urinary disorders) | 2 (2) | 4 (4)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 3 (3)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 8 (9)
Hypotension (Vascular disorders) | 18 (18) | 17 (19)

LIMITATIONS AND CAVEATS:
An interim analysis of 118 subjects was performed by a DRC to assess S. aureus pneumonia rates and the conditional power to detect a statistically significant treatment effect at study completion (354 subjects). The study was terminated for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Primary VAP Prevention Study (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT02940626/Prot_000.pdf
  • Study Protocol: Site-specific VAP Treatment Sub-study (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT02940626/Prot_001.pdf
  • Statistical Analysis Plan: SAP Addendum (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02940626/SAP_002.pdf
  • Statistical Analysis Plan: Primary Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02940626/SAP_003.pdf